CLINICAL TRIAL: NCT06882824
Title: Prevention of HEMOrhagic Risk in Upper MYOmeCTomy by Use of Misoprostol.
Acronym: HEMOMYOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RBHP 2024 GREMEAU
Record Dates: First submitted 2025-01-20; First posted 2025-03-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Myoma;Uterus; Myomectomy; Surgical Blood Loss
Keywords: myomectomy; surgical blood loss; misoprostol
MeSH Terms: conditions — Myofibroma; Blood Loss, Surgical | interventions — Uterine Myomectomy; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment arm with misoprostol (Experimental)
  Interventions: Procedure: myomectomy with misoprostol
- Placebo arm (Placebo Comparator)
  Interventions: Procedure: myomectomy with placebo

INTERVENTIONS:
Procedure: myomectomy with placebo — myomectomy after administration of placebo (control group)
  Arms: Placebo arm
Procedure: myomectomy with misoprostol — myomectomiy after administration of misoprostol 400μg PO (experimental group)
  Arms: treatment arm with misoprostol

SUMMARY:
In France, uterine fibroids or leiomyomas are the most common benign tumour in women of childbearing age.

In 30% of cases, fibroids are symptomatic (menorrhagia, anaemia, pain), in which case surgical management is indicated. This is known as myomectomy, and can be performed by hysteroscopy, laparoscopy (laparoscopy) or laparotomy, depending on the number, size and position of the fibroids.

Intraoperative bleeding is the main surgical difficulty. For this reason, a number of studies have focused on ways of minimizing the risk of bleeding.

A good surgical indication, prevention of anaemia (iron deficiency) and transient occlusion of the uterine arteries during surgery help to reduce this risk. There are also drugs available to reduce intraoperative bleeding, but few studies have been carried out to assess their real effectiveness. One such product is Misoprostol, commonly used in gynecology. Its muscle-contracting properties suggest that it could have a beneficial effect on bleeding during surgery. What's more, this treatment has been used for many years and is reputed to be very well tolerated. The most frequent side effects are digestive, with a risk of abdominal pain in the form of cramps, nausea or vomiting.

The investigators therefore decided to set up the HEMOMYOC study to demonstrate a significant reduction in bleeding during laparotomy or laparoscopic myomectomy after taking oral misoprostol in combination with transient occlusion of the uterine arteries, compared with placebo. It would seem that the ease of use and good tolerance of misoprostol, in combination with transient occlusion of the uterine arteries, could be of real benefit in preventing intraoperative morbidity in myomectomies, whatever the surgical approach. To date, no studies have been carried out in this area.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 43
* Symptomatic myomas (bleeding, pain or infertility)
* Indication for laparoscopic myomectomy Fibroma ≤ 10cm or number ≤ to 4 fibroids
* Indication for myomectomy by laparotomy Fibroma > 10cm, Number > to 4 fibroids
* OTAU possible intraoperatively (Clip on uterine artery and tourniquet placement)
* Speak and understand French
* Affiliated with a social security scheme.

Exclusion Criteria:

* History of major uterine surgery or myomectomy (excluding hysteroscopic myomectomy)
* Allergy to misoprostol and lactose
* Patients with hypersensitivity to misoprostol and/or other prostaglandins or to any of the product's excipients.
* Patients taking aspirin or anti-coagulants
* Patients with haemostasis disorders
* Malnourished patients
* Patients with hepatic or renal insufficiency
* Pregnancy, suspected ectopic pregnancy and breast-feeding women.
* Minors
* Guardianship, curatorship, deprived of liberty, safeguard of justice

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Evaluation of intraoperative blood loss (in milliliters) during myomectomies with OTAU after administration of misoprostol 400μg PO (experimental group) versus placebo (control group) regardless of type of surgery. | during surgery

SECONDARY OUTCOMES:
Evaluate intraoperative blood loss (in milliliters) during myomectomies with OTAU after administration of misoprostol 400μg PO (experimental group) versus placebo (control group) according to surgical technique, laparoscopy and laparotomy. | during surgery
Compare Hemoglobin level (in g/L) between experimental and control groups | between day before surgery and day of surgery
Compare Hemoglobin level (in g/L) between laparotomy and laparoscopy surgery | between day before surgery and day of surgery
Compare between experimental and control groups: Patient age | at inclusion
Compare between laparotomy and laparoscopy: Patient age | at inclusion
Compare between experimental and control groups: Patient BMI | at inclusion
Compare between laparotomy and laparoscopy: Patient BMI | at inclusion
Compare between experimental and control groups: Patient medical history | at inclusion
Compare between laparotomy and laparoscopy: Patient medical history | at inclusion
Compare between experimental and control groups: Patient comorbidities | at inclusion
Compare between laparotomy and laparoscopy: Patient comorbidities | at inclusion
Compare between experimental and control groups: Size of myoma | at inclusion
Compare between laparotomy and laparoscopy: Size of myoma | at inclusion
Compare between experimental and control groups: FIGO classification of myoma | at inclusion
Compare between laparotomy and laparoscopy: FIGO classification of myoma | at inclusion
Compare between experimental and control groups: Number of myoma | at inclusion
Compare between laparotomy and laparoscopy: Number of myoma | at inclusion
Compare between experimental and control groups: Time between tablet intake and incision | day of surgery
Compare between laparotomy and laparoscopy: Time between tablet intake and incision | day of surgery
Compare between experimental and control groups: Total operative time | during surgery
Compare between laparotomy and laparoscopy: Total operative time | during surgery
Compare between experimental and control groups: Transfusion rate in number of RBCs (Red Blood Cells). | during surgery
Compare between laparotomy and laparoscopy: Transfusion rate in number of RBCs (Red Blood Cells). | during surgery
Compare between experimental and control groups: Immediate post-operative complications | up to 8 weeks after surgery
Compare between laparotomy and laparoscopy: Immediate post-operative complications | up to 8 weeks after surgery
Compare between experimental and control groups: Pain assessments at different times: VAS (Visual analogue scale from 0 : no pain to 10 : worst pain) at h+2, h+6 D1 M1 | between 2 hours after surgery until 1 month post-operative
Compare between laparotomy and laparoscopy: Pain assessments at different times: VAS (Visual analogue scale from 0 : no pain to 10 : worst pain) at h+2, h+6 D1 M1 | between 2 hours after surgery until 1 month post-operative
Compare between experimental and control groups: Length of hospital stay after surgery in days | up to one week after surgery
Compare between laparotomy and laparoscopy: Length of hospital stay after surgery in days | up to one week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie GREMEAU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Clermont-Ferrand, France